CLINICAL TRIAL: NCT06811493
Title: Comparison of the Efficacy of One Level and Two Level of Bilateral Thoracic Erector Spinae Plane Block Combined With General Anesthesia in Laparoscopic Bariatric Surgery for Obese Patients: Randomized Controlled Trial.
Brief Title: Comparison of the Efficacy of One Level and Tow Level of Bilateral Thoracic Erector Spinae Plane Block Combined With General Anesthesia in Laparoscopic Bariatric Surgery for Obese Patients: Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Emad Mohamed Ahmed Abdelhafez, lecturer, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MD-407-2024
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Facial Plane Blocks
Keywords: erector spinae plane block, bariatric surgery, obese patients
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- two levels of bilateral thoracic erector spinae plane block (Active Comparator): two level of bilateral thoracic erector spinae plane block combined with general anesthesia in laparoscopic bariatric Surgery for obese patients
  Interventions: Procedure: bilateral thoracic erector spinae plane block combined with general anesthesia in laparoscopic bariatric surgery in obese patients
- one level of bilateral thoracic erector spinae plane block (Active Comparator): one level of bilateral thoracic erector spinae plane block combined with general anesthesia in laparoscopic bariatric Surgery for obese patients
  Interventions: Procedure: bilateral thoracic erector spinae plane block combined with general anesthesia in laparoscopic bariatric surgery in obese patients

INTERVENTIONS:
Procedure: bilateral thoracic erector spinae plane block combined with general anesthesia in laparoscopic bariatric surgery in obese patients — using the in-plane approach, in caudal -to- cephalad direction, through the interfascial plane between the Erector Spinae and the underlying transverse process under strict aseptic precautions until the tip is deep to erector spinae muscle. the block will be performed bilaterally by injecting 60 mL of 0.25% bupivacaine (15 mL into each of four site) into the fascial plane between the deep surface of the Erector Spinae muscle and the bilateral transverse processes of the thoracic vertebrae 5 and 10 (at the most lateral part of the transverse process)

SUMMARY:
comparison of the feasibility and efficacy of the one-level and two-level thoracic ESP block and their effect on intraoperative and postoperative analgesia in bariatric surgeries.

DETAILED DESCRIPTION:
Following approval from Ethics and Research Committee of Anaesthesia Department, Faculty of Medicine, Cairo University; 70 patients fulfilling inclusion criteria will be included in this randomized prospective comparative trial.

A.preoperative:

History will be taken from all patients. Age and then American Society Anaesthesiologists' (ASA) score will be recorded.

Preoperatively patients' laboratory investigations as complete blood picture, coagulation profile, liver and renal functions will be recorded. General examination will be carried out with examination of the back to exclude infection at the injection site and anatomical deformities.

Baseline vital signs will be recorded including non-invasive measurement of systolic, mean, diastolic arterial pressures, and HR and oxygen saturation. After inserting an intravenous (IV) access, the patient will be pre-medicated with metoclopramide in a dose 0.1-0.2 mg/kg.

Patient will be randomly assigned into 1 of 2 groups according to the intervention used whether:

* Group B (Bilevel block) (30 patients): T5 and T10 Erector Spinae block.
* Group O (One level block) (30 patients): T7 Erector Spinae block . Upon arrival to O.R; perioperative monitoring including continuous electrocardiogram (GE-Datex Ohmeda 5 leads ECG cable), pulse oximetry (GE- Datex Ohmeda finger SpO2 sensor), non-invasive arterial blood pressure (GE-Datex Ohmeda NIBP cuff) will be applied.

The block will be performed preoperatively with 1mg midazolam administration intravenous , and 4 cm lidocaine 1% infiltration at each site of block needle prior to the block

In group B, (Bilevel) the block will be performed by the primary investigator . the patient will be placed in the lateral or sitting position . Then, the Erector Spinae block will be given by a high-frequency linear ultrasound transducer of Siemens acuson x300 4.0 - 11.4 MHz ultrasound . It will be sagittally placed against the target vertebral level (T5 transverse process ) (11) in the lateral or sitting position and moved in approximately 3-cm lateral to the spinous process . The Erector Spinae muscle and transverse process will be then identified, and a blunted tip ,100mm, 20-gauge, short bevel needle (Pajunk Sonoplex, Geisingen, Germany) will be advanced, using the in-plane approach, in caudal -to- cephalad direction, through the interfascial plane between the Erector Spinae and the underlying transverse process under strict aseptic precautions until the tip is deep to erector spinae muscle, as evidenced by visible hydro-dissection below the muscle plane, and on injection of 3 ml normal saline to confirm the correct needle tip position and the same technique will be performed at T10 transverse process. The block will be performed bilaterally by injecting 60 mL of 0.25% bupivacaine (15 mL into each of four site) into the fascial plane between the deep surface of the Erector Spinae muscle and the bilateral transverse processes of the thoracic vertebrae 5 and 10 (at the most lateral part of the transverse process) In Group (O) One level The block will be performed bilaterally by injecting 60 mL of 0.25% bupivacaine (30 mL into each side) (12) into the fascial plane between the deep surface of the Erector Spinae muscle and the bilateral transverse processes of the T7 vertebrae by the same technique .

B.intraoperative:

Then, general anaesthesia will be induced in both groups . 1-2 μg/kg fentanyl based on lean body weight (13) with maximum dose of 200 μg and 2 mg/kg propofol will be given based on total body weight (13). Tracheal intubation will be facilitated with 0.5 mg/kg atracurium based on ideal body weight (14).

Anaesthesia will be maintained using isoflurane in oxygen and air. Additional doses of 0.1 mg/kg atracurium will be administrated every 30 minutes. The surgical intervention will be then allowed 20 minutes after finishing the block procedure.

Pressure control volume guarantee ventilation will be adjusted to maintain normocapnia. Anesthesia will be maintained by using 1-1.5% isoflurane in a mixture of oxygen and air (50/50) and atracurium top ups at a dose of 0.1mg/kg every 30 minutes.

All participants will be given 1 gram of intravenous paracetamol every 8 hours Failed block ( increase in HR and mean arterial blood pressure (MABP)>20% from base line with skin incision) will be treated by 1ug /kg of fentanyl as top-up doses and increasing isoflurane concentration in case of inadequate response to fentanyl.

After skin closure, inhalational anesthesia will be discontinued and reversal of muscle relaxation with atropine (0.02 mg/Kg) and neostigmine (0.05 mg/Kg) will be administered intravenous after return of patient's spontaneous breathing. Patients will then be transferred to post anesthesia care unit (PACU) for 60 min to complete recovery and monitoring.

At any time hypotension (defined as a decrease in mean arterial pressure (MAP) >20% from baseline value or systolic arterial pressure (SAP <100 mmHg) will be treated with 5 mg IV bolus ephedrine and repeated every 3 minutes until the hypotension resolved. Bradycardia (defined as a HR less than 15 to 20% of baseline ) will be treated with atropine 0.5 mg IV.(15)

C.postoperative:

In the PACU; VAS will be assessed 30 min after extubation, ketorolac 0.5mg/kg/ 6 hours if VAS score > 3 as first rescue analgesia and nalbuphine as second rescue analgesia 0.1 mg/kg /8 hours as long as the pain score is more than 3\10 ( reassessment to be done after 30 mins of administration of first rescue analgesia ) when the score exceeds 3/10, rescue analgesia in the form of nalbuphine 0.1 mg/Kg will be given. Another dose of nalbuphine 0.1 mg/kg can be given in the PACU if the score still more than 3 after 30 min of the 1st dose with maximum dose of 30 mg every 24 hours.

After discharging from the PACU, the analgesic plan will be intravenous paracetamol one gram every 8 hours , ketorolac 0.5mg/kg/ 6 hours if VAS score > 3 as first rescue analgesia and nalbuphine as second rescue analgesia 0.1 mg/kg /8 hours as long as the pain score is more than 3\10 ( reassessment to be done after 30 mins of administration of first rescue analgesia ).

ELIGIBILITY:
Inclusion Criteria:

* • Patient age ranges 18 to 60 years old

  * Obese patients ; Body mass index(BMI) ≥ 35 - 50 kg/m2
  * American Society of Anesthesiologists (ASA) physical status classes II to III
  * Patients scheduled for laparoscopic bariatric surgery i.e. sleeve gastrectomy and/or Roux-en-Y gastric bypass (RYGB) surgeries

Exclusion Criteria:

* • Refusal of regional block

  * Patients with neurological, psychological disorders or those lacking cooperation
  * Patients scheduled for concomitant laparoscopic cholecystectomy or paraumbilical hernia repair or those with history of previous bariatric surgery or obstructive sleep apnea
  * Patients with anatomic abnormalities at site of injection, skin lesions or wounds at site of proposed needle insertion.
  * Patients with bleeding disorders defined as (INR >1.4) and/ or (platelet count <100,000/µL)
  * Patients with hepatic disease e.g. liver cell failure or hepatic malignancy or hepatic enlargement.
  * Patients who are allergic to amide local anesthetics.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
• visual analog scale (VAS) scores during first 24 hour postoperative | post-operative period at 1 h (hour) , 2 h, 4 h, 8h, 12h,18h and 24 h (hours).
  Pain will be classified as mild (VAS 1-3), moderate (VAS 4-6), and severe (VAS 7-10) .

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No